CLINICAL TRIAL: NCT03211832
Title: Enhancing Evidence-based Diabetes Control Among Local Health Departments
Brief Title: Disseminating Public Health Evidence to Support Prevention and Control of Diabetes Among Local Health Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201705026; 5R01DK109913 (NIH)
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Organizational Support for Evidence-based Public Health
Keywords: Dissemination research; Public health workforce; Evidence-based public health; Public health accreditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will conduct usual public health practice.
- Intervention (Active Comparator): Participating local health departments will help develop and choose several dissemination activities they prefer for their local health department to receive. Dissemination activities may include multi-day in-person training workshops, electronic information exchange modalities, remote technical assistance, and information on ways to enhance organizational climates favorable to evidence-based diabetes and chronic disease prevention and control.
  Interventions: Other: Dissemination of public health knowledge

INTERVENTIONS:
Other: Dissemination of public health knowledge — Participating local health departments will help develop and choose dissemination strategies they prefer for their staff working in and supporting diabetes and chronic disease prevention and control to receive. Dissemination strategies may include multi-day in-person training workshops, electronic information exchange modalities, remote technical assistance, and information on ways to enhance organizational climates favorable to evidence-based diabetes prevention and control.
  Arms: Intervention

SUMMARY:
The purpose of this study is to identify and evaluate dissemination strategies to support the uptake of evidence-based programs and policies (EBPPs) for diabetes prevention and control among local-level public health practitioners. Dissemination strategies such as multi-day in-person training workshops, electronic information exchange modalities, and remote technical assistance are hypothesized to associate with improved access and use of public health evidence and organizational supports for program and policy decision making based on evidence-based public health.

DETAILED DESCRIPTION:
Evidence-based public health approaches to prevent and control diabetes and other chronic diseases have been identified in recent decades, and could have a profound effect on diabetes incidence and quality and length of life of those diagnosed. However, barriers to implement approaches continue because of lack of organizational support, limited resources, competing priorities, and limited skill among the public health workforce. The purpose of this study is to determine effective ways to promote the adoption of evidence based public health practice related to diabetes and chronic disease prevention and control among local health departments (LHDs). This stepped-wedge cluster randomized trial aims to evaluate active dissemination strategies on local-level public health practitioners to increase adoption and use of evidence-based programs and policies for diabetes and chronic disease prevention and control among LHDs in Missouri. Twelve LHDs will be recruited and randomly assigned to one of three groups that cross over from usual practice to receive the intervention (dissemination) strategies at 8-month intervals; the intervention duration for groups ranges from 8 to 24 months. LHD staff and the university-based study team are jointly identifying, refining and selecting dissemination strategies. Intervention strategies may include multi-day in-person training workshops, electronic information exchange modalities, and remote technical assistance. Evaluation methods include surveys at baseline and at each 8-month interval, abstraction of LHD chronic disease prevention program plans and progress reports, and social network analysis.

ELIGIBILITY:
Inclusion Criteria:

* Local Health Departments (LHDs, cluster) in the state of Missouri and corresponding public health workforce (individuals within cluster); screenings.

Exclusion Criteria:

* LHDs that have less than 5 employees working in or supporting diabetes or chronic disease control, which includes program areas of diabetes prevention and management, obesity prevention, physical activity, nutrition, cardiovascular health, and cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross C Brownson, PhD, Principal Investigator — Prevention Research Center in St. Louis, Brown School, Washington University in St. Louis, Division of Public Health Sciences, Department of Surgery and Alvin J. Siteman Cancer Center, Washington University School of Medicine
Locations (1):
- Prevention Research Center, Brown School, Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parks RG, Tabak RG, Allen P, Baker EA, Stamatakis KA, Poehler AR, Yan Y, Chin MH, Harris JK, Dobbins M, Brownson RC. Enhancing evidence-based diabetes and chronic disease control among local health departments: a multi-phase dissemination study with a stepped-wedge cluster randomized trial component. Implement Sci. 2017 Oct 18;12(1):122. doi: 10.1186/s13012-017-0650-4. PMID 29047384
- [Result] Jacob RR, Parks RG, Allen P, Mazzucca S, Yan Y, Kang S, Dekker D, Brownson RC. How to "Start Small and Just Keep Moving Forward": Mixed Methods Results From a Stepped-Wedge Trial to Support Evidence-Based Processes in Local Health Departments. Front Public Health. 2022 Apr 28;10:853791. doi: 10.3389/fpubh.2022.853791. eCollection 2022. PMID 35570955
- See also: Click here for more information about this study: Adoption and Implementation of evidence to Mobilize Local Health — https://prcstl.wustl.edu/items/aim-local-health/
- See also: Protocol paper — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5648488/
- See also: Results paper — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9096224/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 local public health departments were recruited into the study in 3 groups. Once a health department agreed to participate, health department managers provided employee lists for self-report survey invitations.
Pre-assignment Details: Each group of 4 health departments crossed over into intervention at different times.
  In the stepped-wedge design, at baseline, surveys from all 12 health departments were analyzed as control surveys. Once a health department had crossed over into intervention, all remaining surveys of that health department's employees were analyzed as intervention surveys. At the last survey data collection, all surveys were analyzed as intervention surveys.
Units Other Than Participants: Health departments/agencies
Groups:
- Group 1 - Control (2 Months), Then Intervention (24 Months): While in control status, the health departments will conduct usual public health practice.
  During Intervention, each health department will help develop and choose several dissemination activities they prefer for their local health department to receive. Dissemination activities may include multi-day in-person training workshops, electronic information exchange modalities, remote technical assistance, and information on ways to enhance organizational climates favorable to evidence-based diabetes and chronic disease prevention and control.
  Dissemination of public health knowledge: Participating local health departments will help develop and choose dissemination strategies they prefer for their staff working in and supporting diabetes and chronic disease prevention and control to receive. Dissemination strategies may include multi-day in-person training workshops, electronic information exchange modalities, remote technical assistance, and information on ways to enhance organizational climates favorable to evidence-based diabetes prevention and control.
- Group 2 - Control (10 Months), Then Intervention (16 Months); Group 3 - Control (18 Months), Then Intervention (8 Months): While in control status, the health department conducted usual public health practice.
  Intervention began with a multi-day training in evidence-based decision making. Then each health department selected and helped develop intra-organizational procedures, policies, and additional activities to embed evidence-based decision making into day-to-day public health practice.
Period: Overall Study
Arm/Group | Group 1 - Control (2 Months), Then Intervention (24 Months) | Group 2 - Control (10 Months), Then Intervention (16 Months) | Group 3 - Control (18 Months), Then Intervention (8 Months)
Started (Baseline Survey. All participants were employees at participating local health departments.) | 78; 4 Health departments/agencies (In Group 1, 78 health department employees agreed to participate and completed the baseline survey.) | 85; 4 Health departments/agencies (In Group 2, 85 health department employees agreed to participate and completed the baseline survey.) | 66; 4 Health departments/agencies (In Group 3, 66 health department employees agreed to participate and completed the baseline survey.)
Survey Time 2 (At Survey Time 2, 37 health department employees were added to replace those no longer working at the agency.) | 83; 4 Health departments/agencies (Group 1 was in intervention status at Survey Time 2 and so Group 1 participant surveys were analyzed as intervention. At Survey Time 2, 8 health department employees were added to replace those no longer working at the health department. In Group 1, 83 unique individuals completed the Time 2 survey.) | 87; 4 Health departments/agencies (At Survey Time 2, Group 2 was still in control status. At Survey Time 2, 19 health department employees were added to replace those no longer working at the health department. A total of 87 unique individual health department employees in Group 2 completed the Time 2 survey.) | 63; 4 Health departments/agencies (At Survey Time 2, Group 3 was still in control status. Ten health department employees were added to replace those no longer at the agency. In Group 3, 63 unique individuals completed the survey at Time 2.)
Survey Time 3 (More unique health department employee participants were again added (27 due to employee turnover and 15 to better reflect Group 2 health department units involved in the intervention).) | 70; 4 Health departments/agencies (In Group 1, 6 health department employees were added to replace employees no longer at the health department. At Survey Time 3, 70 unique individuals completed the survey.) | 112; 4 Health departments/agencies (Groups 1 and 2 were in intervention status at Survey Time 3 and so their employee participant surveys were analyzed as intervention. Ten health department employees were added at Survey Time 3 to replace those no longer with the agency and 15 more were added to better reflect participating units within the health departments. At Survey Time 3, 112 unique individuals completed the survey in Group 2.) | 55; 4 Health departments/agencies (Group 3 was still in control status at Survey Time 3. Eleven health department employees were added at Survey Time 3 to replace those no longer working at the agency.)
Survey Time 4 (At Survey Time 4, all groups were in Intervention status. At Survey Time 4, 23 health department employees were added to replace those no longer working at the health departments.) | 70; 4 Health departments/agencies (At Survey Time 4, 7 health department employees were added to replace those no longer with the health departments.70 unique individuals completed the Time 4 survey.) | 97; 4 Health departments/agencies (At Survey Time 4, 10 health department employees were added to replace some of those no longer with the health departments.) | 60; 4 Health departments/agencies (At Survey Time 4, 6 health department employees were added to replace those no longer with the agency.)
Completed | 42; 4 Health departments/agencies (In the stepped wedge design, all groups were in intervention at the last data collection. 227 unique individuals completed self-report surveys at the end of the study, but only a portion of these had completed the baseline survey. A total of 331 unique individuals completed the survey at one or more time points.) | 33; 4 Health departments/agencies | 32; 4 Health departments/agencies
Not Completed | 36; 0 Health departments/agencies | 52; 0 Health departments/agencies | 34; 0 Health departments/agencies
Not completed — No longer with agency | 32 | 49 | 30
Not completed — Declined survey | 3 | 3 | 2
Not completed — Not available during data collection | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The unit of analysis is surveys. In the stepped-wedge design, analyses were conducted on the completed surveys, not unique individuals, since all individual health department employee survey participants were controls at the beginning and crossed over to intervention before the last survey data collection.
Units Other Than Participants: completed surveys
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (completed surveys) | 433 | 489 | 922
Age, Customized [Number; unit: completed surveys]
  18-29 years | 103 | 92 | 195
  30-39 years | 111 | 127 | 238
  40-49 years | 88 | 100 | 188
  50-59 years | 88 | 116 | 204
  >=60 years | 42 | 52 | 94
  Not reported | 1 | 2 | 3
Sex: Female, Male [Count of Units; unit: completed surveys]
  Female | 356 | 411 | 767
  Male | 77 | 78 | 155
Race/Ethnicity, Customized [Count of Units; unit: completed surveys] — Race/Ethnicity Not Collected. Population: Race/Ethnicity was not collected, therefore the number analyzed of zero is different from the overall number of surveys analyzed for the other measures.
  completed surveys
    number analyzed (completed surveys) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: completed surveys]
  United States | 433 | 489 | 922

OUTCOME MEASURES:

1. Primary Outcome: Evidence-based Decision Making (EBDM) Competencies
Description: Survey participants were asked to rate the perceived importance of each of 10 skills pertinent to evidence-based decision making on an 11-point ordered scale (possible values 0 not at all important to 10 very important for each skill), and to rate the perceived availability in the agency of each of the same skills from 0-10 (0 not at all available to 10 very available). A skill gap was calculated for each skill as perceived importance minus perceived availability (possible values -10 to +10 for each skill). An overall EBDM skill gap was created by taking the average across all 10 skill gaps (possible values -10 to +10). Higher scores indicate a worse outcome.
  Skill items: community assessment; quantifying the issue; prioritization; action planning; adapting interventions; evaluation designs; quantitative evaluation; qualitative evaluation; economic evaluation; and communicating evidence to decision-makers. A definition for each was provided that started with the word "understand".
Time Frame: 24 months post baseline
Population: The unit of analysis is completed surveys due to the stepped-wedge design and having a different set of survey participants at each of the 4 survey time points. All baseline surveys were analyzed as control; at T4 all surveys were analyzed as intervention. Survey participants were health department employees. Due to staff turnover, some had left the agency between each data collection period and others hired, so additional health department staff were invited at Survey T2, T3, and T4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: completed surveys
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (completed surveys) | 433 | 489
score on a scale | 2.05 [1.87 to 2.23] | 1.98 [1.82 to 2.13]

2. Primary Outcome: Evidence-based Intervention Score
Description: Self-reported number of evidence-based chronic disease prevention interventions implemented by the local health department from a pre-populated list of 8 evidence-based interventions to prevent diabetes and other chronic diseases (possible score 0 to 8). Higher score indicates a better outcome.
Time Frame: 24 months post baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: completed surveys
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (completed surveys) | 433 | 489
units on a scale | 4.84 [4.61 to 5.07] | 4.58 [4.36 to 4.80]

3. Primary Outcome: Awareness of Culture Supportive of EBDM
Description: Self-report Likert scale items measure personal awareness of opportunities to learn about and apply EBDM among local level chronic disease control public health practitioners. Each item is measured on a 7-point Likert scale from 1 strongly disagree to 7 strongly agree. A summary score was created as an average of the items within the domain. Possible scores 1 to 7. Higher scores mean a better outcome.
  The items were: a) I am provided the time to identify evidence-based programs and practices; b) My direct supervisor recognizes the value of management practices that facilitate evidence-based decision-making; c) My work group/division offers employees opportunities to attend evidence-based-decision making trainings; and d) Top leadership in my agency (e.g., director, assistant directors) recognizes the value of evidence-based decision-making.
Time Frame: 24 months post baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: completed surveys
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (completed surveys) | 433 | 489
score on a scale | 5.34 [5.22 to 5.47] | 5.43 [5.31 to 5.54]

4. Primary Outcome: Capacity and Expectations for Evidence-based Decision Making (EBDM)
Description: Self-report Likert scale items assess perceived supervisory expectations for EBDM use and perceived work unit/division capacity to carry out EBDM. Each item is measured on a 7-point Likert scale from 1 strongly disagree to 7 strongly agree. A summary score was created as an average of the items (possible scores 1 to 7). Higher scores mean a better outcome.
  Items: a) I use EBDMin my work; b) My direct supervisor expects me to use evidence-based decision making; c) My performance is partially evaluated on how well I use evidence-based decision making in my work; d) My work group/division currently has the resources (e.g. staff, facilities, partners) to support application of evidence-based decision making; e) The staff in my work group/division has the necessary skills to carry out evidence-based decision making; f) The majority of my work group/division's external partners support use of EBDM; and g) Top leadership in my agency encourages use of EBDM.
Time Frame: 24 months post baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: completed surveys
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (completed surveys) | 433 | 489
score on a scale | 5.22 [5.11 to 5.33] | 5.24 [5.14 to 5.35]

5. Primary Outcome: Resource Availability
Description: Self-report Likert scale items measured perceived work unit's resource availability for evidence-based decision making. Each item is measured on a 7-point Likert scale from 1 strongly disagree to 7 strongly agree. A summary score was created as an average of the items. Possible scores 1 to 7. Higher scores mean a better outcome.
  The items in the scale were: a) Informational resources (e.g. academic journals, guidelines, and toolkits) are available to my work group/division to promote the use of evidence-based decision making; b) My work group/division engages a diverse external network of partners that share resources to facilitate evidence-based decision making; and c) Stable funding is available for evidence-based decision making.
Time Frame: 24 months post baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: completed surveys
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (completed surveys) | 433 | 489
score on a scale | 4.46 [4.32 to 4.60] | 4.47 [4.35 to 4.60]

6. Primary Outcome: Evaluation Capacity of Work Unit
Description: Self-report Likert scale of work unit's support of community needs assessment, utilization of evaluation for pre and post program implementation as well as for dissemination purposes. Each item is measured on a 7-point Likert scale from 1 strongly disagree to 7 strongly agree. A summary score was created as an average of the items within the domain. Possible scores 1 to 7. Higher scores mean a better outcome.
  Items: a) My work group/division supports community needs assessments to ensure that evidence-based decision-making approaches continue to meet community needs; b) My work group/division plans for evaluation of interventions prior to implementation; c) My work group/division uses evaluation data to monitor and improve interventions; and d) My work group/division distributes intervention evaluation findings to other organizations that can use our findings.
Time Frame: 24 months post baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: completed surveys
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (completed surveys) | 433 | 489
score on a scale | 5.23 [5.10 to 5.33] | 5.19 [5.07 to 5.31]

7. Primary Outcome: EBDM Climate Cultivation
Description: Self-report Likert scale assessing perceived health department culture supportive of EBDM, information sharing and participatory decision making. Each item is measured on a 7-point Likert scale from 1 strongly disagree to 7 strongly agree. A summary score was created as an average of the items within the domain. Possible scores 1 to 7. Higher scores mean a better outcome.
  Items: a) My work group/division has access to evidence-based decision making information that is relevant to community needs; b) When decisions are made within my work group/division, program staff members are asked for input; c) Information is widely shared in my work group/division so that everyone who makes decisions has access to all available knowledge; d) My agency is committed to hiring people with relevant training or experience in public health core disciplines (e.g., epidemiology, health education, environmental health); and e) My agency has a culture that supports the processes necessary for EBDM.
Time Frame: 24 months post baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: completed surveys
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (completed surveys) | 433 | 489
score on a scale | 5.21 [5.08 to 5.34] | 5.26 [5.14 to 5.37]

8. Primary Outcome: Partnerships to Support EBDM
Description: Self-report Likert scale items assess perceived importance of partnering across sectors to share resources and address population health issues. Each item is measured on a 7-point Likert scale from 1 strongly disagree to 7 strongly agree. A summary score was created as an average of the items within the domain. Possible scores 1 to 7. Higher scores mean a better outcome.
  Items: a) Our collaborative partnerships have missions that align with my agency; b) It is important to my agency to have partners who share resources (money, staff time, space, materials); c) It is important to my agency to have partners in health care to address population health issues; and d) It is important to my agency to have partners in other sectors (outside of health) to address population health issues
Time Frame: 24 months post baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: completed surveys
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (completed surveys) | 433 | 489
score on a scale | 5.94 [5.86 to 6.03] | 5.91 [5.83 to 6.00]

9. Secondary Outcome: Inter-agency Connectedness
Description: The average number of links per agency is the measure of connectedness with other agencies that is reported here. The measure is from a separate self-report social network survey.
Time Frame: 24 months post baseline
Population: Agencies with completed social network surveys at baseline when all health departments were in control status and at the end of the study when all health departments were in the intervention.
Measure: Mean (Standard Deviation); unit: Agencies
Units Other Than Participants: Agencies
Arm/Group | Control | Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (Agencies) | 224 | 261
Agencies | 6.8 (1.7) | 8.5 (2.7)

ADVERSE EVENTS:
Description: Clinical adverse event data were not collected because there were no study outcomes involving a health behavior, a disease or health condition, a symptom, or health status. Outcomes were perceived capacity for and organizational supports for use of evidence-based decision making among public health department employees.
  The main risk to participants was loss of confidentiality of survey response, which was monitored. No losses of confidentiality were found by or reported to the study team.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The stepped-wedge design allowed all 12 health departments to participate in intervention but completing surveys at 4 time points was a burden to employees. Due to staff turnover, we added new employees at each time point, and lost others due to no longer working at the health department. Responses to the quantitative survey were self-reported, which introduces the possibility of response bias. Response rates dropped at the last data collection in spring 2020 during LHD pandemic efforts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT03211832/Prot_SAP_000.pdf